CLINICAL TRIAL: NCT01333358
Title: Phase III A Prospective, Longitudinal, Rater-blinded Single-arm Study to Evaluate Alemtuzumab as an Effective Treatment in Stabilizing Overall Neurocognitive Function in RRMS Subjects at Specified Timepoints
Brief Title: Evaluating Alemtuzumab as a Treatment in Stabilizing Neurocognitive Function In Relapsing Remitting Multiple Sclerosis Patients
Acronym: CAMA-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Texas Neurology Consultants (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Central Texas Neurology Consultants, Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 111746
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing; remitting
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab 12mg given intravenously each day for five days and again twelve months later for an additional three days
  Other Names: Campath Mabcampath

SUMMARY:
The main purpose of this research study is to investigate how well a medicine (alemtuzumab) works in treating MS-related cognitive problems (e.g., attention, memory, speed of thinking). This study will include 30 subjects from six research sites.

Alemtuzumab is approved and sold under the brand names Campath and MabCampath to treat some types of leukemia. As a leukemia treatment, it is given more often and at much higher doses than in this study.

DETAILED DESCRIPTION:
The current proposal is to conduct a study using a battery of neuropsychological tests capable of detecting the broad range of cognitive difficulties associated with relapsing remitting multiple sclerosis. This study will compare cognitive functioning over time of patients receiving alemtuzumab. The study will also compare the change in cognitive functioning over time to that of relapsing remitting multiple sclerosis patients receiving interferon beta-1a and normal controls enrolled in a parallel study conducted by Wilken et al.To evaluate cognitive effects of alemtuzumab, the investigators will perform neurological exams and brain scans and will administer questionnaires to measure the severity of multiple sclerosis, how well subjects are functioning, how they are feeling, and to find out about what other medical visits subjects may have had during the study. Neurological testing in this study will require the subject to perform relatively simple tasks to evaluate their multiple sclerosis. These tasks include a five hundred meter walk, a timed twenty five foot walk, a nine hole peg test, an eye exam, and a test requiring you to add small numbers in your head quickly. The brain scans will involve Magnetic Resonance Imaging and are painless, except for injection of a contrast agent called gadolinium, which is necessary to detect areas in the brain where their MS may be currently active. Magnetic Resonance Imaging is widely used to diagnose and assess patients with multiple sclerosis. All patients will be required to return to their study site every 3 months for assessments and testing. In addition, safety-related blood tests will be performed at least monthly. If their blood test results become abnormal, they may have to have blood tests taken more frequently, in some cases weekly, until test results improve. Monthly blood tests should be performed at your study site, but if subjects are unable to return to the study site for the blood testing, they may be able to use a local laboratory.

Participation in this study should last at least 4 years and possibly longer.

Subjects receiving alemtuzumab, will need to have blood tests every month for at least 3 years after your last dose of alemtuzumab. Therefore, you will need to undergo monthly blood tests for a total of about 4 years. If your test results become abnormal, you may have to have blood tests more frequently, in some cases weekly, until your test results improve.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. Age 18 to 55 years old (inclusive) as of the date the ICF is signed
3. Diagnosis of MS per McDonald criteria (2005 update).
4. Onset of MS symptoms (as determined by a neurologist, at present or retrospectively) within 10 years of the date the ICF is signed
5. EDSS score 0.0 to 5.0 (inclusive) at Screening
6. ≥ 2 MS attacks (first episode or relapse) occurring in the 24 months prior to the date the ICF is signed, with ≥ 1 attack in the 12 months prior to the date the ICF is signed, with objective neurological signs confirmed by a physician, nurse practitioner, or other sponsor-approved health-care provider. The objective signs may be identified retrospectively.
7. ≥ 1 MS attack (relapse) during treatment with a beta interferon therapy or glatiramer acetate after having been on that therapy for ≥ 6 months within 10 years of the date the ICF is signed
8. MRI scan demonstrating white matter lesions attributable to MS and meeting at least 1 of the following criteria, as determined by the neurologist or a radiologist

   * ≥ 9 T2 lesions at least 3 mm in any axis
   * a gadolinium-enhancing lesion at least 3 mm in any axis plus > 1 brain T2 lesions
   * a spinal cord lesion consistent with MS plus > 1 brain T2 lesions
9. Corrected vision of subjects must be no worse than 20/50.
10. Participants must have at least 10 years of education.
11. Participants must be capable of writing and pressing the buttons on a computer mouse.
12. Participants must be capable of understanding and following all test instructions.

Exclusion Criteria:

Patients will be excluded from enrollment in this study if they meet any of the following criteria:

1. Previous treatment with alemtuzumab
2. Current participation in another clinical study or previous participation in CAMMS323
3. Treatment with natalizumab, methotrexate, azathioprine, or cyclosporine in the past 6 months. Patients who received one of these medications more than 6 months before the date the ICF is signed may be eligible for study entry if approval is granted by the sponsor
4. Previous treatment with mitoxantrone, cyclophosphamide, cladribine, rituximab or any other immunosuppressant or cytotoxic therapy (other than steroids)
5. Previous treatment with any investigational medication (drug has not been approved at any dose or for any indication) unless prior approval is granted by the sponsor and the patient completes any required washout. Use of an investigational medication that was subsequently licensed and nonstandard use of a licensed medication (eg, using a dose other than the dose that is stated in the licensed product labeling or using a licensed therapy for an alternative indication) is not exclusionary. Prior treatment with herbal medications or nutritional supplements is also permitted.
6. Any progressive form of MS
7. History of malignancy, except basal skin cell carcinoma
8. Any disability acquired from trauma or another illness that, in the opinion of the Investigator, could interfere with evaluation of disability due to MS
9. Previous hypersensitivity reaction to any immunoglobulin product
10. Known allergy or intolerance to interferon beta, human albumin, or mannitol
11. Intolerance of pulsed corticosteroids, especially a history of steroid psychosis
12. Inability to self-administer SC injections or receive SC injections from caregiver
13. Inability to undergo MRI with gadolinium administration
14. Confirmed platelet count < the lower limit of normal (LLN) of the evaluating laboratory at Screening or documented at <100,000/μL within the past year on a sample without platelet clumping
15. Absolute neutrophil count < LLN at Screening; if abnormal cell count returns to within normal limits, eligibility may be reassessed
16. Known bleeding disorder (eg, dysfibrinogenemia, factor IX deficiency, hemophilia, Von Willebrand's disease, disseminated intravascular coagulation [DIC], fibrinogen deficiency, clotting factor deficiency)
17. Seropositivity for human immunodeficiency virus (HIV)
18. Significant autoimmune disease including but not limited to: immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders, vasculitis, inflammatory bowel disease, severe psoriasis.
19. Active infection, eg, deep-tissue infection, that the Investigator considers sufficiently serious to preclude study participation
20. In the Investigator's opinion, is at high risk for infection (eg, indwelling catheter, dysphagia with aspiration, decubitus ulcer, history of prior aspiration pneumonia or recurrent urinary tract infection)
21. Latent tuberculosis unless effective anti-tuberculosis therapy has been completed, or active tuberculosis.
22. Infection with hepatitis C virus
23. Past or present hepatitis B infection (positive hepatitis B serology)
24. Of childbearing potential with a positive serum pregnancy test, pregnant, or lactating
25. Unwilling to agree to use a reliable and acceptable contraceptive method throughout the study period (fertile patients only). Reliable and effective contraceptive method(s) include: intrauterine device (IUD), hormonal based contraception, surgical sterilization, abstinence, or double-barrier contraception (condom and occlusive cap (diaphragm or cervical cap with spermicide).
26. Major psychiatric disorder that is not adequately controlled by treatment
27. Epileptic seizures that are not adequately controlled by treatment
28. Major systemic disease or other illness that would, in the opinion of the Investigator, compromise patient safety or interfere with the interpretation of study results, e.g., current peptic ulcer disease, or other conditions that may predispose to hemorrhage
29. Medical, psychiatric, cognitive, or other conditions that, in the Investigator's opinion, compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study
30. Prior history of invasive fungal infections
31. Cervical high risk human papillomavirus (HPV) positivity or abnormal cervical cytology other than abnormal squamous cells of undetermined significance (ASCUS). The patient may be eligible after the condition has resolved (e.g., follow-up HPV test is negative or cervical abnormality has been effectively treated).
32. Any other illness or infection (latent or active) that, in the Investigator's opinion, could be exacerbated by either study medication
33. Any hepatic or renal function value grade 2 or higher at Screening, with the exception of hyperbilirubinemia due to Gilbert's syndrome, unless, in the Investigator's opinion, the abnormality is due to a condition that has resolved (eg, recent interferon treatment subsequently discontinued) and levels return to within normal limits. See Table below, drawn from the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE), published 09 August 2006.

    * Hepatic
    * Bilirubin > 1.5 × ULN
    * SGOT/AST > 2.5 × ULN
    * SGPT/ALT > 2.5 × ULN
    * Alkaline phosphatase > 2.5 × ULN
    * Renal
    * Creatinine > 1.5 × ULN
34. Participants with upper extremity dysfunction which prohibits them from using a computer mouse.
35. Participants who are colorblind.
36. Participants with current alcohol/substance abuse.
37. Participants taking medications with notable adverse CNS effects such as excessive sedation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The primary study objective is to demonstrate whether treatment with alemtuzumab is effective in stabilizing overall neurocognitive functioning in relapsing-remitting multiple sclerosis over time. | Four years
  To determine the rate of change in cognitive scores for RRMS participants taking alemtuzumab over time. The data from participants in this trial will be compared to data from normal controls and RRMS patients receiving Rebif® in a parallel trial conducted by Wilken et al (in preparation).

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Fox, MD,PhD, Principal Investigator — Central Texas Neurology Consultants